CLINICAL TRIAL: NCT06556329
Title: Using Artificial Intelligence (AI) - Enhanced Social Robots to Improve Children's Healthcare Experiences
Brief Title: Canada-UK AI Study
Acronym: Canada-UK AI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00097697
Record Dates: First submitted 2024-07-11; First posted 2024-08-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Social Robots for Procedural Distress
Keywords: artificial intelligence; social robotics; procedural distress; child pain; children
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: The intervention arm will have a socially assistive, artificially enhanced robot presence during an intravenous insertion procedure; the standard of care arm will follow standard procedures that are practiced clinically.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Control) (No Intervention): This arm will include topical anesthetic as well as a combination of parental support, child life services and/or healthcare provider support, at the discretion of the treating team and family.
- Robot (Intervention) (Experimental): This arm will include the addition of robot distraction to current departmental standard of care. Distraction will include interaction with a socially intelligent, autonomous humanoid robot, the development of which will be informed by the other work packages.
  Interventions: Other: Robot (Intervention)

INTERVENTIONS:
Other: Robot (Intervention) — The research team will bring a socially assistive, artificially-enhanced robot during intravenous insertion procedures.
  Arms: Robot (Intervention)

SUMMARY:
Children experience pain and distress in clinical settings every day. The negative consequences of unaddressed pain can be both short-term (e.g. fear, distress, inability to perform procedures) and long-term (e.g. needle phobia, anxiety).

In previous small studies, a humanoid robot has been used to deliver cognitive-behavioural therapy during needle procedures. The results of these early studies have been positive, showing high acceptance among children as well as promising initial clinical results. However, these studies all had critical technical limitations: the robot was remotely operated and used purely scripted behaviour with limited Artificial Intelligence support. This reduced the potential to offer personalized support to children. In this project, the study team aims to address this limitation by developing and evaluating a clinically relevant and responsive artificial intelligence-enhanced social robot.

DETAILED DESCRIPTION:
PURPOSE:

The study team aims to develop and evaluate an artificial intelligence-enhanced socially intelligent robot designed to alleviate children's distress and pain in a clinical setting.

HYPOTHESIS:

The study team believes that interaction with a robust, adaptive, socially intelligent robot can effectively distract children during painful clinical procedures, thereby reducing pain and distress.

JUSTIFICATION:

A recent review examined eight studies where a robot was used to reduce children's pain and distress: overall, while the results seem promising, there is also a need for improved methodology and measures to draw conclusions. In particular, the authors suggest more effective interventions could be created by ensuring that healthcare experts and engineers collaborate from the start, and that user and family partners contribute to a user-centred design process. Our proposed work includes such family input and research team collaboration. Previous reviews have also identified an urgent need to increase the autonomy of the robots to improve their robustness and adaptability. Our project will aim to address this by developing and evaluating a responsive AI-enhanced social robot.

In addition, as AI systems such as robots grow more pervasive in daily life, understanding the impact of such systems on society has become ever more crucial. For social robots, in particular, an important consideration is determining the social role that the robot should play, as well as an ethical and appropriate means of making clear the capabilities of the robot.

METHODS:

* Months 24-36; University of Alberta, University of Toronto
* The goal is to conduct a clinical trial of the robot system developed in Study Design: This randomized controlled superiority trial will consist of two arms: (1) The Standard of Care (Control) Arm will include topical anesthetic cream as well as a combination of parental support, child life services and/or healthcare provider support, at the discretion of the treating team and family. (2) The Robot (Intervention) Arm will include the addition of robot distraction to current departmental standard of care. Distraction will include interaction with a socially intelligent, autonomous humanoid robot, the development of which will be informed by the earlier stages of this study (co-design and usability phases).

Primary Objective: Our primary objective of is to compare the reduction of pain and distress with the use of distraction (via the robot intervention) versus current standard of care in children aged 5 to 11 years who are undergoing intravenous insertion (IVI).

Secondary Objectives: The secondary objectives are (a) to compare the reduction of fear in the robot intervention versus standard of care arms; (b) to compare the reduction of parental/caregiver anxiety with their child's use of robot intervention versus standard of care; (c) to compare child, parental/caregiver and nurse satisfaction with the procedure in the intervention versus standard of care arms; (d) to examine the association between parental/caregiver anxiety and child outcomes (ie. pain, distress, fear); (e) to assess children's degree of engagement with the socially intelligent, autonomous humanoid robot; and (f) to assess the ethical needs and issues related to interaction with a socially intelligent, autonomous humanoid robot.

Data Collection: Research Assistants (RAs) will screen the electronic emergency department trackboard and communicate with on-site clinical staff to identify potentially eligible patients. For children flagged as requiring an IVI the RA will further assess eligibility, and acquire informed consent/ assent as appropriate. The RA will then gather baseline demographic/ history information and access a secure Research Electronic Data Capture (REDCap) randomization tool to determine the child's group assignment (ie. either Robot intervention or Control group).

Approximately five minutes prior to the start of the procedure (defined as cleaning of the IV site), the RA will begin the video recording and collect pre-procedure pain, fear and parental anxiety measures. For children randomized to the intervention group, the RA will bring in the robot and explain how to interact with it. The clinical nurse will then insert the IV following standard institutional protocols. For children randomized to the intervention group, the RA will bring in the robot and explain how to interact with it. The clinical nurse will then insert the IV following standard institutional protocols. Immediately following the first attempt at IVI (regardless of success), the RA will repeat the pain, fear and parental anxiety measures. Within 5-10 minutes of the procedure, satisfaction and acceptability questionnaires will be completed with the child, parent/ caregiver and the clinical nurse. Video recording will conclude 5 minutes after the procedure and only one attempt will be recorded, regardless of success of the IVI. Video recording will allow for coding of OSBD-R distress scores at a later time. Visit details will be collected from the child's medical chart.

Setting and Sample: The study team plans to recruit 85-90 patients in total. Patients will be recruited from the emergency departments of the Stollery Children's Hospital (Edmonton) and SickKids (Toronto).

PLAN FOR DATA ANALYSIS (clinical data):

Statistical analyses will be conducted using statistical software Statisical Analysis Software (SAS) (version 9; SAS Institute, Cary, North Carolina). Baseline variables will be described using appropriate summary statistics. For pain during the procedure, the mean (or median, if appropriate) scores will be compared between the two groups using independent samples t-tests (normal distribution) or Mann-Whitney U-tests (skewed). For Observational Scale of Behavioral Distress-Revised (OSBD-R), a change score (during procedure minus pre-procedure) will be calculated for each child, and the mean change scores will be compared between study groups (Mann-Whitney U test). Multiple linear regression analyses will be conducted with distress as the response variable, baseline pain and group indicators as explanatory variables, and possible effect modifiers (i.e. age, sex). Intention-to-treat approach will be used. The significance level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. child aged 5-11 years
2. requires IVI
3. will receive topical anesthetic for IVI

Exclusion Criteria:

1. medically unstable (CTAS 1, requiring immediate IV insertion)
2. unconscious or not fully alert
3. visual or auditory impairments
4. neurocognitive delays or mental health issues precluding safe interaction with the robot intervention
5. sensory impairment to pain (ex. spina bifida)
6. parental or child language barrier precluding the ability to understand and complete study assessments, in the absence of a native language translator
7. not accompanied by legal guardian
8. previous enrolment in this clinical trial or in the co-design or usability studies
9. other reason at the discretion of the clinical staff

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Self-reported pain level | Scores will be taken 5 minutes before intravenous intervention and immediately after intravenous insertion (approximately 3-4 minutes post-procedure)
  Compare the reduction of pain with the use of distraction (via the robot intervention) versus current standard of care in children aged 5 to 11 years who are undergoing IVI.
  The investigators will use the following scales:
  - Pain score: Faces Pain Scale-Revised (score: 0-10; 10 being worst pain)
Self-reported distress level | Scores will be taken 5 minutes before intravenous intervention and immediately after intravenous insertion (approximately 3-4 minutes post-procedure)
  Compare the reduction of pain and distress with the use of distraction (via the robot intervention) versus current standard of care in children aged 5 to 11 years who are undergoing IVI.
  The investigators will use the following scales:
  - Distress score: Numerical rating scale (score: 0-10; 10 being most distressed)

SECONDARY OUTCOMES:
Self-reported fear level | Scores will be taken 5 minutes before intravenous intervention and immediately after intravenous insertion (approximately 3-4 minutes post-procedure)
  To compare the reduction of fear in the robot intervention versus standard of care arms.
  The investigators will use the following scale:
  - Children's Fear Scale (score: 0-4; 4 being the most scared)
Parental/caregiver anxiety | Scores will be taken 5 minutes before intravenous intervention and immediately after intravenous insertion (approximately 3-4 minutes post-procedure)
  To compare the reduction of parental/caregiver anxiety with their child's use of robot intervention versus standard of care.
  The investigators will use the following scale:
  - State Trait Anxiety Inventory, Form Y-1 (STAI) (score: sum 20-80; higher score = more anxious)
Satisfaction with procedure | Outcome will be measured immediately after intravenous insertion (approximately 3-4 minutes post-procedure)
  To compare child, parental/caregiver and nurse satisfaction with the procedure in the intervention versus standard of care arms.
  The investigators will use the following scales:
  - 5-point Likert scales asking questions on satisfaction (overall IV insertion, pain management, agreeability to use same distraction tool)
Engagement | Outcome will be measured immediately after intravenous insertion (approximately 3-4 minutes post-procedure)
  To assess children's degree of engagement with the socially intelligent, autonomous humanoid robot.
  - Assessed by the standard Robot Semantic Attribute Scale (18-item scale); score: sum 18-126; higher score = better engagement

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets and open-source software will also be made available via providing the research team's contact information on our publication.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: July 01, 2025 for 10 years thereafter.
Access Criteria: Interested research teams will be required to provide proof of research ethics approval